CLINICAL TRIAL: NCT00185367
Title: A Multi-center, Double-blind, Double-dummy, Controlled, Randomized Study to Evaluate Cycle Control and Safety of a Four Phasic Oral Contraceptive (SH T00658ID) in Comparison to an Oral Contraceptive Containing Ethinylestradiol and Levonorgestrel (SH D 593 B) in Healthy Female Volunteers Aged Between 18 and 50 Years.
Brief Title: Comparative Cycle Control Europe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 90883; EudraCT: 2004-001613-34; 304004
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K)
- Arm 2 (Active Comparator)
  Interventions: Drug: SH D 593 B (Miranova)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K) — 7 cycles each consisting of 28 days (no tablet-free intervals); Day 1-2: 3.0 mg EV; Day 3-7: 2.0 mg EV + 2.0 mg DNG; Day 8-24: 2.0 mg EV + 3.0 mg DNG; Day 25-26: 1.0 mg EV; Day 27-28: placebo;In addition SH D 593 B (Miranova) matching placebo
  Arms: Arm 1
Drug: SH D 593 B (Miranova) — 7 cycles each consisting of 28 days (no tablet-free intervals); Day 1-21: 0.02 mg EE + 0.10 mg LNG; Day 22-28: placebo; In addition EV/DNG (Qlaira, BAY86-5027, SH T00658K) matching placebo
  Arms: Arm 2

SUMMARY:
The aim of this study is to evaluate bleeding pattern, cycle control, and safety of this new four-phasic oral contraceptive in comparison to a reference OC.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers aged between 18 and 50 years requiring contraception

Exclusion Criteria:

* Pregnancy or lactation
* Any conditions that might interfere with the outcome as well as all contraindications for OC use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 798 (Actual)
Dates: Start 2005-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bleeding pattern | 7 treatment cycles each consisting of 28 days
Number of unintended pregnancies | 7 treatment cycles each consisting of 28 days and follow-up period of 14 days

SECONDARY OUTCOMES:
Adverse event collection | 7 treatment cycles each consisting of 28 days and follow-up period of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (34):
- Czechia (5):
  - Soukroma gynekologicka ambulance, Fulnek
  - Soukroma gynekologicka ambulance, Pilsen
  - Provozorna Gynekologicka ordinace Dr. Tesar, Prague
  - Femina Sana s.r.o, Prague
  - Soukroma gynekologicka ambulance, Zábřeh nad Odrou
- France (10):
  - Dr. Jocelyne Nataf-Maurin, Brignoles
  - Dr. Marie-Helene Malbranche-Aupecle, Dijon
  - Centre Hospitalier de l Estuaire, Honfleur
  - Dr. Annette Mercier, Morlaix
  - Clinique d Occitanie, Muret
  - Centre Medical du Val de Loire, Nevers
  - Dr. Anne-Isabelle Richet, Paris
  - Cabinet medical, Quetigny
  - Dr. Gwendoline Servan, Tarare
  - Dr. Aliette Siboni-Frisch, Toulouse
- Germany (19):
  - Frauenarztpraxis Dr. Buchberger, Neubiberg, Bavaria
  - Praxis Hr. Dr. R. Kuett, Nuremberg, Bavaria
  - Praxis Dr. Larbig, Fulda, Hesse
  - Praxis Fr. Dr. J. Schmidt-Pich, Hanover, Lower Saxony
  - Praxis Fr. Dr. A. Münzberger, Döbeln, Saxony
  - Praxis Fr. Dr. K. Kopprasch, Dresden, Saxony
  - Praxis Fr. R. Hellmich, Dresden, Saxony
  - Frauenarztpraxis Dr. Bernd Pittner, Leipzig, Saxony
  - Praxis Fr. Dr. C. Burgkhardt, Leipzig, Saxony
  - Frauenarztpraxis Dr. Wetzel, Blankenburg, Saxony-Anhalt
  - Frauenarztpraxis Dipl. med. Michael Stellmacher, Burg, Saxony-Anhalt
  - Praxis Fr. Dr. A. Braune, Magdeburg, Saxony-Anhalt
  - Praxis Hr. Prof. Dr. H.-J. Ahrendt, Magdeburg, Saxony-Anhalt
  - Frauenarztpraxis Hr. Dr. H. Lindecke, Berlin, State of Berlin
  - Praxis Fr. Dr. B. Heuberger, Berlin, State of Berlin
  - Praxis Hr. Dr. Karl-Heinz Belling, Berlin, State of Berlin
  - Frauenarztpraxis Hr. Dr. B. Hamann, Berlin, State of Berlin
  - Praxis Hr. R. Wähnert, Gera, Thuringia
  - Praxis Fr. Dr. A.Mönch-Hering, Kahla, Thuringia

REFERENCES:
- [Derived] Ahrendt HJ, Makalova D, Parke S, Mellinger U, Mansour D. Bleeding pattern and cycle control with an estradiol-based oral contraceptive: a seven-cycle, randomized comparative trial of estradiol valerate/dienogest and ethinyl estradiol/levonorgestrel. Contraception. 2009 Nov;80(5):436-44. doi: 10.1016/j.contraception.2009.03.018. Epub 2009 May 13. PMID 19835717